CLINICAL TRIAL: NCT00813917
Title: Varenicline for the Treatment of Smokeless Tobacco Use
Brief Title: Varenicline for the Treatment of Smokeless Tobacco
Acronym: CHANCHEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Jon Ebbert, MD, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-005359; CA132621-01A1
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Results first posted 2011-09-09 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- varenicline (Active Comparator)
  Interventions: Drug: varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: varenicline — 12 weeks of varenicline 1 mg by mouth twice per day
  Other Names: Chantix
  Arms: varenicline
Drug: placebo — 12 weeks of placebo (double blinded) by mouth twice per day
  Other Names: Chantix placebo
  Arms: Placebo

SUMMARY:
Varenicline (Chantix™, Pfizer) is a novel selective nicotinic receptor partial agonist with specificity for the α4β2 nicotine acetylcholine receptor that has demonstrated remarkable efficacy for increasing long-term tobacco abstinence rates in cigarette smokers. The novel mechanism of action of varenicline potentially circumvents the limitations of using nicotine replacement therapy or bupropion pharmacotherapy in ST users. The overall goal of this line of research is to develop effective pharmacologic treatments for ST users to increase long-term (≥ 6 months) abstinence rates. The central hypothesis of this application is that varenicline is efficacious for the treatment of ST users.

DETAILED DESCRIPTION:
In the United States, approximately 7.7 million individuals older than 12 years of age report current (past month) use of smokeless tobacco (ST). ST use has been associated with oral and extra-oral cancer as well as cardiovascular and cerebrovascular disease. To date, no pharmacotherapies have been shown to increase long-term (≥ 6 months) abstinence rates in ST users. Novel pharmacotherapies that decrease withdrawal symptoms and nicotine self-administration need to be tested in ST users. Varenicline (Chantix™, Pfizer) is a novel selective nicotinic receptor partial agonist with specificity for the α4β2 nicotine acetylcholine receptor that has demonstrated remarkable efficacy for increasing long-term tobacco abstinence rates in cigarette smokers. The novel mechanism of action of varenicline potentially circumvents the limitations of using nicotine replacement therapy or bupropion pharmacotherapy in ST users. The overall goal of this line of research is to develop effective pharmacologic treatments for ST users to increase long-term (≥ 6 months) abstinence rates. The central hypothesis of this application is that varenicline is efficacious for the treatment of ST users. To evaluate this hypothesis, we will conduct a pilot study to obtain preliminary estimates of efficacy of 12-weeks of varenicline for increasing the prolonged and point prevalence tobacco abstinence rates at 12 weeks (end-of-treatment) in ST users. We will also evaluate the effect of varenicline on nicotine withdrawal symptoms and tobacco craving. If the results are promising, we will plan for a multicenter, randomized, double-blinded, placebo-controlled clinical trial with the Oregon Research Institute in Eugene, OR, to investigate the efficacy of varenicline to increase long-term (≥ 6 months) abstinence rates in ST users.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to participate if they:

1. Are at least 18 years of age
2. Have used ST daily for the past 12 months (regular user)
3. Identify ST as their primary tobacco product
4. Are in general good health (determined by medical history and screening physical examination)
5. Has provided written informed consent to participate
6. Are able to participate in all aspects of the study

Exclusion Criteria:

Individuals will be excluded from study participation if they:

1. Are currently (in previous 30 days) using other behavioral or pharmacologic tobacco cessation programs (i.e., behavioral therapy, nicotine replacement therapy, clonidine, bupropion SR, or doxepin)
2. Have self-reported current, untreated depression or a Beck Depression Inventory (BDI-II) Score of ≥ 20
3. Have, as defined by the C-SSRS (Columbia-Suicide Severity Rating Scale);current non-specific suicidal thoughts, or have a lifetime history of a suicidal attempt (defined as "potentially self-injurious act committed with at least some wish to die, as a result of act.")
4. History of psychosis or bipolar disorder
5. Are currently pregnant or lactating or is of childbearing potential and not willing to use any form of contraception
6. Have another member of their household already participating in this study
7. Are allergic to varenicline
8. Describe having a medical history of:

   * Unstable angina
   * Myocardial infarction within the past 3 months
   * Cardiac dysrhythmia other than medication-controlled atrial fibrillation or PSVT
   * Medically-treated or untreated hypertension with BP ≥ 200 systolic OR ≥ 100 diastolic
   * Have other medical or psychiatric conditions that would exclude the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon O. Ebbert, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Nicotine Research Program, Rochester, Minnesota, United States

REFERENCES:
- [Result] Ebbert JO, Croghan IT, Severson HH, Schroeder DR, Hays JT. A pilot study of the efficacy of varenicline for the treatment of smokeless tobacco users in Midwestern United States. Nicotine Tob Res. 2011 Sep;13(9):820-6. doi: 10.1093/ntr/ntr078. Epub 2011 Apr 18. PMID 21504885
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 4/13/09 and completed on 08/16/10. Interested subjects who passed a phone pre-screen were seen at a medical clinic (Mayo Clinic in Rochester, MN and Franciscan Skemp Medical Center in Lacrosse, WI) for consenting and additional study procedures to determine eligibility.
Groups:
- Varenicline: varenicline-1mg/day for 12 weeks
- Placebo: nonactive lookalike pill per day for 12 weeks
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 38 | 38
Completed | 32 | 32
Not Completed | 6 | 6
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 36 | 74
  >=65 years | 0 | 2 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 41.0 (12.4) | 40.7 (10.1) | 40.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 38 | 38 | 76
smokeless tobacco quantity [Mean (Standard Deviation); unit: cans per week] — Amount of smokeless tobacco used per week
  cans per week | 4.0 (3.5) | 3.2 (2.0) | 3.6 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence All Tobacco Abstinence
Description: 7-day point prevalence all tobacco abstinence at week 12 (end of treatment)confirmed by urine cotinine less than 50ng/ml
Time Frame: 12 weeks - end of treatment
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 38 | 38
participants | 21 | 16
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Data were compared between treatment groups using Chi Square test; Test type: Superiority or Other; p = 0.126, Chi-squared — For this randomized phase II we used a one sided test with a false positive(type I error)rate of 0.20 to assess whether additional studies of the experimental arm are warranted; 1 sided

ADVERSE EVENTS:
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 15/38 | 5/38
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=38) | Placebo (N=38)
Nausea (Gastrointestinal disorders) | 9 | 0
sleep disturbance (General disorders) | 7 | 3
vivid dreams (General disorders) | 3 | 1
headache (General disorders) | 1 | 1
confusion (General disorders) | 0 | 1
constipation (Gastrointestinal disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 0 | 1
dizziness (General disorders) | 1 | 0
hives (General disorders) | 1 | 0
irritability (General disorders) | 1 | 0
mood disturbance (General disorders) | 0 | 1
restlessness (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No